CLINICAL TRIAL: NCT00526097
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of 4 Weeks Treatment With Bisacodyl (Dulcolax) Tablets 10mg Administered Orally, Once Daily, in Patients With Functional Constipation.
Brief Title: Dulcolax vs Placebo in Functional Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 122.56; EUDRACT 2007-001991-34
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Results first posted 2010-08-06 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2013-12

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Bisacodyl

ARMS (2):
- Bisacodyl 5 mg x 2 once daily (Experimental): patient to receive two enteric-coated tablets containing 5 mg bisacodyl
  Interventions: Drug: Bisacodyl 10 mg
- Placebo (Placebo Comparator): patient to receive two placebo-to-match enteric-coated tablets 5 mg bisacodyl
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bisacodyl 10 mg — 2 x 5 mg bisacodyl once daily
  Arms: Bisacodyl 5 mg x 2 once daily
Drug: Placebo — Placebo-to-match bisacodyl 10 mg (2 x 5 mg) once daily
  Arms: Placebo

SUMMARY:
The objective of the study was to compare the efficacy and safety of 4 weeks treatment with bisacodyl (Dulcolax) tablets 10 mg to placebo in patients with functional constipation. In addition, the effect of treatment on quality of life and general health status was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, aged 18 and above
2. Suffering from functional constipation, according to their medical history, as defined by the Rome III diagnostic criteria , i.e.:Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.

   1. Must include 2 or more of the following::

      * straining during at least 25% of the defecations
      * lumpy or hard stools in at least 25% of the defecations
      * sensation of incomplete evacuation for at least 25% of the defecations
      * sensation of anorectal obstruction/blockade for at least 25% of the defecations
      * manual manoeuvres to facilitate at least 25% of the defecations (e.g. digital evacuation, support of the pelvic floor)
      * fewer than 3 defecations per week
   2. Loose stools are rarely present without the use of laxatives
   3. There are insufficient criteria for irritable bowel syndrome (IBS)
3. Able and willing to complete a daily e-diary
4. Able and willing to use the trial rescue medication
5. Signed and dated written informed consent prior to enrolment into the study in accordance with GCP and local legislation

   At Visit 2, patients must comply with the following additional inclusion criteria to be eligible for entry into the treatment phase:
6. Functional constipation is confirmed by e-diary data at the end of the baseline period:

   a. An average of less than 3 CSBMs per week, together with at least one of the following symptoms occurring at least 25% of the time:
   * straining
   * incomplete evacuation
   * lumpy or hard stools (i.e. type 1 or type 2 stools)
7. Compliant with the use of the e-diary throughout the baseline period (compliance is defined as completing 80% of the evening reports)
8. Compliant with the use of rescue medication throughout the baseline period. Compliance is defined as follows:

   * rescue medication may be used if there has not been a bowel movement for more than 72 hrs rescue medication may not be used on either day -1 or on the day of randomisation (day 1)

Exclusion Criteria:

1. Eating disorders such as anorexia nervosa and bulimia, as a cause of excessive use of laxatives
2. Patients whose constipation is caused by primary organic disease of the colon or pelvic floor
3. Patients with metabolic disorders, neurological disorders, severe or psychiatric disorders, or any other significant disease or intercurrent illness (e.g. abdominal/gastrointestinal surgery) that, in the Investigators opinion, would interfere with participation in the trial
4. Patients with restricted mobility (e.g. wheelchair bound, or bed-ridden) that, in the Investigators opinion, would interfere with participation in the trial
5. Patients with a known hypersensitivity to bisacodyl or any other ingredient in the study medication
6. Patients with ileus, intestinal obstruction, acute surgical abdominal conditions (such as acute appendicitis and acute inflammatory bowel diseases), or severe dehydration
7. Patients with anal fissures or ulcerative proctitis with mucosal damage
8. Patients with known clinically significant abnormal electrolyte values
9. Patients whose concomitant therapy includes an opioid medication (e.g. morphine, codeine)
10. Constipation which, in the Investigators opinion, is caused by medication (e.g. anticholinergics)
11. Patients who are not willing to discontinue the use of prohibited concomitant therapy
12. Pre-menopausal women who:

    1. are nursing (breast-feeding) or who are pregnant OR
    2. who are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study. Acceptable methods of birth control include:

       * transdermal patch
       * intra-uterine devices/systems (IUDs/IUSs)
       * oral, implantable or injectable contraceptives
       * sexual abstinence
       * sterilisation or a vasectomised partner
13. Participation in another trial with an investigational product with 1 month of enrolment into this study
14. Drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (27):
- United Kingdom (27):
  - 122.56.44032 Boehringer Ingelheim Investigational Site, Addlestone
  - 122.56.44018 Boehringer Ingelheim Investigational Site, Ash Vale, Aldershot
  - 122.56.44029 Boehringer Ingelheim Investigational Site, Ashford
  - 122.56.44023 Boehringer Ingelheim Investigational Site, Atherstone
  - 122.56.44011 Boehringer Ingelheim Investigational Site, Bedworth
  - 122.56.44009 Boehringer Ingelheim Investigational Site, Bennetthorpe, Doncaster
  - 122.56.44025 Boehringer Ingelheim Investigational Site, Bexhill-on-Sea
  - 122.56.44012 Boehringer Ingelheim Investigational Site, Blackpool
  - 122.56.44024 Boehringer Ingelheim Investigational Site, Burbage
  - 122.56.44003 Boehringer Ingelheim Investigational Site, Cardiff
  - 122.56.44017 Boehringer Ingelheim Investigational Site, Chesterfield
  - 122.56.44014 Boehringer Ingelheim Investigational Site, Chippenham
  - 122.56.44006 Boehringer Ingelheim Investigational Site, Chorley
  - 122.56.44033 Boehringer Ingelheim Investigational Site, Dundee
  - 122.56.44002 Boehringer Ingelheim Investigational Site, Edgbaston, Birmingham
  - 122.56.44004 Boehringer Ingelheim Investigational Site, Glasgow
  - 122.56.44007 Boehringer Ingelheim Investigational Site, Liverpool
  - 122.56.44005 Boehringer Ingelheim Investigational Site, Manchester
  - 122.56.44010 Boehringer Ingelheim Investigational Site, Midsomer Norton
  - 122.56.44021 Boehringer Ingelheim Investigational Site, Newtonabbey
  - 122.56.44022 Boehringer Ingelheim Investigational Site, Paignton
  - 122.56.44020 Boehringer Ingelheim Investigational Site, Royal Leamington Spa
  - 122.56.44001 Boehringer Ingelheim Investigational Site, Slough
  - 122.56.44026 Boehringer Ingelheim Investigational Site, Sunbury-on-Thames
  - 122.56.44019 Boehringer Ingelheim Investigational Site, Swindon
  - 122.56.44015 Boehringer Ingelheim Investigational Site, Warminster
  - 122.56.44008 Boehringer Ingelheim Investigational Site, Wolverhampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were partly recruited by commercial research centers and partly by general practitioners.
Pre-assignment Details: Participants were randomised into the treatment period only, when functional constipation and compliance with rescue medication were confirmed by eDiary data in the two-weeks baseline period without study medication.
Groups:
- Placebo: Two bisacodyl-matching 5 mg placebo tablets once daily
- Bisacodyl: Two bisacodyl 5 mg tablets once daily
Period: Overall Study
Arm/Group | Placebo | Bisacodyl
Started | 121 (Started: Participant was randomised and took at least one dose of randomised study medication) | 247 (Started: Participant was randomised and took at least one dose of randomised study medication)
Completed | 106 (Completed: Participant without premature discontinuation in the randomised treatment period) | 191 (Completed: Participant without premature discontinuation in the randomised treatment period)
Not Completed | 15 | 56
Not completed — Adverse Event | 6 | 44
Not completed — Protocol Violation | 4 | 10
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bisacodyl | Total
Number analyzed (Participants) | 121 | 247 | 368
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (15.1) | 55.8 (15.9) | 55.4 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 179 | 275
  Male | 25 | 68 | 93
Baseline assessment regarding the bothersomeness with abdominal bloating [Number; unit: Participants] — Baseline assessment was made at the end of the last week of the baseline period without study medication using a 5-point ordinal VRS: 0 (Not at all bothersome) to 4 (A very great deal bothersome)
  Participants
    Not at all bothersome | 12 | 21 | 33
    Hardly bothersome | 20 | 33 | 53
    Moderately bothersome | 40 | 85 | 125
    A good deal bothersome | 36 | 60 | 96
    A very great deal bothersome | 12 | 47 | 59
    Missing assessment | 1 | 1 | 2
Baseline assessment regarding the bothersomeness with abdominal discomfort [Number; unit: Participants] — Baseline assessment was made at the end of the last week of the baseline period without study medication using a 5-point ordinal VRS: 0 (Not at all bothersome) to 4 (A very great deal bothersome)
  Participants
    Not at all bothersome | 14 | 26 | 40
    Hardly bothersome | 22 | 40 | 62
    Moderately bothersome | 47 | 91 | 138
    A good deal bothersome | 31 | 64 | 95
    A very great deal bothersome | 6 | 25 | 31
    Missing assessment | 1 | 1 | 2
Baseline assessment regarding the bothersomeness with constipation [Number; unit: Participants] — Baseline assessment was made at the end of the last week of the baseline period without study medication using a 5-point ordinal VRS: 0 (Not at all bothersome) to 4 (A very great deal bothersome)
  Participants
    Not at all bothersome | 6 | 15 | 21
    Hardly bothersome | 5 | 19 | 24
    Moderately bothersome | 57 | 91 | 148
    A good deal bothersome | 41 | 88 | 129
    A very great deal bothersome | 11 | 33 | 44
    Missing assessment | 1 | 1 | 2
Baseline assessment regarding the overall satisfaction with bowel habits [Number; unit: Participants] — Baseline assessment was made at the end of the last week of the baseline period without study medication using a 5-point ordinal verbal rating scale (VRS): 0 (A very great deal satisfied) to 4 (Not at all satisfied)
  Participants
    A very great deal satisfied | 3 | 10 | 13
    A good deal satisfied | 3 | 9 | 12
    Moderately satisfied | 41 | 74 | 115
    Hardly satisfied | 44 | 93 | 137
    Not at all satisfied | 29 | 60 | 89
    Missing assessment | 1 | 1 | 2
Baseline for dimension 'Bodily pain (BP)' of the SF-36 QoL scale [Mean (Standard Deviation); unit: Score on a scale] — The dimension is a sum of 2 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
  Score on a scale | 68.5 (24.3) | 67.5 (26.0) | 67.8 (25.4)
Baseline for dimension 'General health (GH)' of the SF-36 QoL scale [Mean (Standard Deviation); unit: Score on a scale] — The dimension is a sum of 5 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health. (Placebo: N=119, Bisacodyl: N=245)
  Score on a scale | 68.0 (21.1) | 69.9 (20.6) | 69.3 (20.7)
Baseline for dimension 'Mental health (MH)' of the SF-36 QoL scale [Mean (Standard Deviation); unit: Score on a scale] — The dimension is a sum of 5 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
  Score on a scale | 74.2 (18.0) | 77.0 (16.8) | 76.1 (17.2)
Baseline for dimension 'Physical functioning (PF)' of the SF-36v2™ (SF-36) Quality of Life (QoL) [Mean (Standard Deviation); unit: Score on a scale] — The dimension is a sum of 10 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
  Score on a scale | 79.2 (24.3) | 80.1 (24.6) | 79.8 (24.5)
Baseline for dimension 'Role limitation due to emotional problems (RE)' of the SF-36 QoL scale [Mean (Standard Deviation); unit: Score on a scale] — The dimension is a sum of 3 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
  Score on a scale | 82.7 (24.7) | 86.3 (22.3) | 85.1 (23.1)
Baseline for dimension 'Role limitation due to physical problems (RP)' of the SF-36 QoL scale [Mean (Standard Deviation); unit: Score on a scale] — The dimension is a sum of 4 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
  Score on a scale | 79.7 (25.2) | 80.6 (25.6) | 80.3 (25.5)
Baseline for dimension 'Social functioning (SF)' of the SF-36 QoL scale [Mean (Standard Deviation); unit: Score on a scale] — The dimension is a sum of 2 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
  Score on a scale | 83.4 (21.6) | 86.0 (20.9) | 85.1 (21.2)
Baseline for dimension 'Vitality (VT)' of the SF-36 QoL scale [Mean (Standard Deviation); unit: Score on a scale] — The dimension is a sum of 4 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
  Score on a scale | 55.7 (20.2) | 58.9 (21.0) | 57.9 (20.8)
Baseline for the Mental Component Scale (MCS) of the SF-36 QoL scale [Mean (Standard Deviation); unit: Score on a scale] — The MCS is a summary scale of the dimensions vitality, social functioning, role-emotional, and mental health. The component scale is norm-based to a standard population. A higher score indicates a better health. (Placebo: N=119, Bisacodyl: N=245)
  Score on a scale | 49.0 (11.0) | 51.1 (9.8) | 50.4 (10.3)
Baseline for the Physical Component Scale (PCS) of the SF-36 QoL scale [Mean (Standard Deviation); unit: Score on a scale] — The PCS is a summary scale of the subscales physical functioning, role-physical, bodily pain, and general health. The component scale is norm-based to a standard population. A higher score indicates a better health. (Placebo: N=119, Bisacodyl: N=245)
  Score on a scale | 48.7 (9.4) | 48.3 (9.8) | 48.5 (9.7)
Baseline mean score for constipation symptom 'Sensation of incomplete evacuation' [Mean (Standard Deviation); unit: Score on a scale] — The score on a 2-point ordinal verbal rating scale from 0 (no) to 1 (yes) specifying patient's symptom assessment associated with each bowel movement was averaged over the day and then averaged over the days in the last week of the baseline period without study medication (Placebo: N=120, Bisacodyl: N=240).
  Score on a scale | 0.7 (0.3) | 0.7 (0.3) | 0.7 (0.3)
Baseline mean score for constipation symptom 'Manual manoeuvre' [Mean (Standard Deviation); unit: Score on a scale] — The score on a 2-point ordinal verbal rating scale from 0 (no) to 1 (yes) specifying patient's symptom assessment associated with each bowel movement was averaged over the day and then averaged over the days in the last week of the baseline period without study medication (Placebo: N=116, Bisacodyl: N=231).
  Score on a scale | 0.2 (0.4) | 0.2 (0.3) | 0.2 (0.3)
Baseline mean score for constipation symptom 'Anorectal obstructions/blockade' [Mean (Standard Deviation); unit: Score on a scale] — The score on a 5-point ordinal verbal rating scale from 0 (absent) to 4 (very severe) specifying patient's symptom assessment associated with each bowel movement was averaged over the day and then averaged over the days in the last week of the baseline period without study medication. (Placebo: N=116, Bisacodyl: N=231)
  Score on a scale | 1.2 (1.0) | 1.2 (1.0) | 1.2 (1.0)
Baseline mean score for constipation symptom 'Stool quality' [Mean (Standard Deviation); unit: Score on a scale] — The score on the 7-point Bristol Stool Form Scale from Type 1 (hard, lumpy stool) to Type 7 (watery stool) specifying patient's symptom assessment associated with each bowel movement was averaged over the day and then averaged over the days in the last week of the baseline period without study medication. (Placebo: N=116, Bisacodyl: N=231)
  Score on a scale | 2.4 (1.2) | 2.5 (1.3) | 2.4 (1.3)
Baseline mean score for constipation symptom 'Straining' [Mean (Standard Deviation); unit: Score on a scale] — The score on a 5-point ordinal verbal rating scale from 0 (absent) to 4 (very severe) specifying patient's symptom assessment associated with each bowel movement was averaged over the day and then averaged over the days in the last week of the baseline period without study medication. (Placebo: N=116, Bisacodyl: N=231)
  Score on a scale | 1.9 (0.9) | 1.8 (0.8) | 1.9 (0.8)
Baseline number of Complete Spontaneous Bowel Movements (CSBMs) [Mean (Standard Deviation); unit: CSBMs per week] — Complete Spontaneous Bowel Movement (CSBM): complete non-rescue medication-induced BM; Baseline number of CSBMs is defined by the number of CSBMs during the last week of the baseline period without study medication
  CSBMs per week | 1.0 (1.1) | 1.1 (1.2) | 1.1 (1.2)
Baseline number of Spontaneous Bowel Movements (SBMs) [Mean (Standard Deviation); unit: SBMs per week] — Spontaneous BM (SBM): non-rescue medication-induced BM; Baseline number of SBMs is defined by the number of SBMs during the last week of the baseline period without study medication
  SBMs per week | 4.2 (2.6) | 4.4 (3.9) | 4.3 (3.6)
Baseline overall score (OSC) of PAC-QoL [Mean (Standard Deviation); unit: Score on a scale] — The PAC-QoL is a 28-item (5-point Likert scale ranging from 0 (none of the time or not at all) to 4 (all of the time or extremely). Single item scores are inverted, if applicable, to ensure that a lower score indicates a better QoL (Placebo: N=119, Bisacodyl: N=245)
  Score on a scale | 1.8 (0.6) | 1.8 (0.7) | 1.8 (0.7)
Baseline subscore 'Physical discomfort (PHD)' of PAC-QoL [Mean (Standard Deviation); unit: Score on a scale] — The PAC-QoL is a 28-item (5-point Likert scale ranging from 0 (none of the time or not at all) to 4 (all of the time or extremely). Single item scores are inverted, if applicable, to ensure that a lower score indicates a better QoL (Placebo: N=120, Bisacodyl: N=245)
  Score on a scale | 1.9 (0.8) | 2.0 (0.9) | 2.0 (0.9)
Baseline subscore 'Psychosocial discomfort (PSD)' of PAC-QoL [Mean (Standard Deviation); unit: Score on a scale] — The PAC-QoL is a 28-item (5-point Likert scale ranging from 0 (none of the time or not at all) to 4 (all of the time or extremely). Single item scores are inverted, if applicable, to ensure that a lower score indicates a better QoL (Placebo: N=121, Bisacodyl: N=245)
  Score on a scale | 0.8 (0.8) | 0.9 (0.8) | 0.9 (0.8)
Baseline subscore 'Satisfaction (SAT)' of PAC-QoL [Mean (Standard Deviation); unit: Score on a scale] — The PAC-QoL is a 28-item (5-point Likert scale ranging from 0 (none of the time or not at all) to 4 (all of the time or extremely). Single item scores are inverted, if applicable, to ensure that a lower score indicates a better QoL (Placebo: N=120, Bisacodyl: N=245)
  Score on a scale | 3.0 (0.7) | 2.8 (0.8) | 2.9 (0.8)
Baseline subscore'Worries and concerns (WCC)' of Patient Assessment of Constipation-QoL(PAC-QoL) [Mean (Standard Deviation); unit: Score on a scale] — The PAC-QoL is a 28-item (5-point Likert scale ranging from 0 (none of the time or not at all) to 4 (all of the time or extremely). Single item scores are inverted, if applicable, to ensure that a lower score indicates a better QoL (Placebo: N=121, Bisacodyl: N=245)
  Score on a scale | 1.4 (0.8) | 1.5 (0.9) | 1.4 (0.9)
Baseline value for chloride (normalized value) [Mean (Standard Deviation); unit: mmol/L] — Normalized value: the reported laboratory value is converted by linear transformation to a preferred unit and then linear-transformed with respect to the standard reference range (Placebo: N=120, Bisacodyl: N=245)
  mmol/L | 104.0 (2.33) | 103.7 (2.85) | 103.8 (2.69)
Baseline value for potassium (normalized value) [Mean (Standard Deviation); unit: mmol/L] — Normalized value: the reported laboratory value is converted by linear transformation to a preferred unit and then linear-transformed with respect to the standard reference range (Placebo: N=120, Bisacodyl: N=244)
  mmol/L | 4.2 (0.33) | 4.2 (0.33) | 4.2 (0.33)
Baseline value for sodium (normalized value) [Mean (Standard Deviation); unit: mmol/L] — Normalized value: the reported laboratory value is converted by linear transformation to a preferred unit and then linear-transformed with respect to the standard reference range (Placebo: N=120, Bisacodyl: N=245)
  mmol/L | 139.5 (2.13) | 139.3 (2.30) | 139.4 (2.24)

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Complete Spontaneous Bowel Movements (CSBMs) Per Week Over the 4 Weeks Treatment Period
Description: A Complete Spontaneous Bowel Movement (CSBM) is a complete non-rescue medication-induced stool.
  The number of CSBMs in each of the 4 weeks was divided by the number of days where data were available in this week, multiplied by 7 and rounded off to the next integer. The sum of the resulting numbers were divided by the number of weeks with data.
Time Frame: 4 Weeks
Population: Full Analysis Set (FAS): All randomised patients, who recorded at least one dose of trial medication in the eDiary and provided any data for the primary outcome measure
Measure: Least Squares Mean (Standard Error); unit: CSBMs per week
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
CSBMs per week | 1.9 (0.34) | 5.2 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — Treatment differences (Bisacodyl - Placebo) were estimated by reference to the adjusted least squares mean differences and the corresponding 95% confidence intervals (CIs); Mean Difference (Final Values) = 3.3, 95% CI [2.6 to 4.0], Standard Error of Mean 0.36 — Means are adjusted for center effects and baseline value

2. Secondary Outcome: Number of CSBMs at Week 1
Description: The number of CSBMs at week 1 was divided by the number of days where data were available in this week, multiplied by 7 and rounded off to the next integer.
Time Frame: Week 1 in treatment period
Population: Patients from FAS (= All randomised patients, who recorded at least one dose of trial medication in the eDiary and provided any data for the primary outcome measure), who provided data for the underlying outcome measure
Measure: Least Squares Mean (Standard Error); unit: CSBMs per week
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
CSBMs per week | 2.0 (0.40) | 6.3 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.3, 95% CI [3.5 to 5.2], Standard Error of Mean 0.42 — Means are adjusted for center effects and baseline value

3. Secondary Outcome: Number of CSBMs at Week 2
Description: The number of CSBMs at week 2 was divided by the number of days where data were available in this week, multiplied by 7 and rounded off to the next integer.
Time Frame: Week 2 in treatment period
Population: Patients from FAS ( = All randomised patients, who recorded at least one dose of trial medication in the eDiary and provided any data for the primary outcome measure), who provided data for the underlying outcome measure
Measure: Least Squares Mean (Standard Error); unit: CSBMs per week
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 115 | 229
CSBMs per week | 1.4 (0.41) | 4.9 (0.33)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.5, 95% CI [2.7 to 4.3], Standard Error of Mean 0.43 — Means are adjusted for center effects and baseline value

4. Secondary Outcome: Number of CSBMs at Week 3
Description: The number of CSBMs at week 3 was divided by the number of days where data were available in this week, multiplied by 7 and rounded off to the next integer.
Time Frame: Week 3 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: CSBMs per week
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 113 | 213
CSBMs per week | 1.8 (0.38) | 4.6 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.8, 95% CI [2.0 to 3.6], Standard Error of Mean 0.39 — Means are adjusted for center effects and baseline value

5. Secondary Outcome: Number of CSBMs at Week 4
Description: The number of CSBMs at week 4 was divided by the number of days where data were available in this week, multiplied by 7 and rounded off to the next integer.
Time Frame: Week 4 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: CSBMs per week
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 196
CSBMs per week | 1.7 (0.42) | 4.3 (0.35)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.6, 95% CI [1.8 to 3.4], Standard Error of Mean 0.43 — Means are adjusted for center effects and baseline value

6. Secondary Outcome: Mean Number of SBMs Per Week Over the 4 Weeks Treatment Period
Description: A Spontaneous Bowel Movement (SBM) is a non-rescue medication-induced stool. The number of SBMs in each of the 4 weeks was divided by the number of days where data were available in this week, multiplied by 7 and rounded off to the next integer. The sum of the resulting numbers were divided by the number of weeks with data.
Time Frame: 4 Weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: SBMs per week
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
SBMs per week | 5.1 (0.41) | 10.0 (0.33)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.9, 95% CI [4.1 to 5.8], Standard Error of Mean 0.43 — Means are adjusted for center effects and baseline value

7. Secondary Outcome: Number of SBMs at Week 1
Description: The number of SBMs at week 1 was divided by the number of days where data were available in this week, multiplied by 7 and rounded off to the next integer.
Time Frame: Week 1 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: SBMs per week
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
SBMs per week | 5.3 (0.46) | 12.1 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.7, 95% CI [5.8 to 7.7], Standard Error of Mean 0.49 — Means are adjusted for center effects and baseline value

8. Secondary Outcome: Number of SBMs at Week 2
Description: The number of SBMs at week 2 was divided by the number of days where data were available in this week, multiplied by 7 and rounded off to the next integer.
Time Frame: Week 2 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: SBMs per week
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 115 | 229
SBMs per week | 4.9 (0.44) | 9.6 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.7, 95% CI [3.8 to 5.6], Standard Error of Mean 0.46 — Means are adjusted for center effects and baseline value

9. Secondary Outcome: Number of SBMs at Week 3
Description: The number of SBMs at week 3 was divided by the number of days where data were available in this week, multiplied by 7 and rounded off to the next integer.
Time Frame: Week 3 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: SBMs per week
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 113 | 213
SBMs per week | 4.8 (0.44) | 8.6 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.8, 95% CI [2.9 to 4.7], Standard Error of Mean 0.45 — Means are adjusted for center effects and baseline value

10. Secondary Outcome: Number of SBMs at Week 4
Description: The number of SBMs at week 4 was divided by the number of days where data were available in this week, multiplied by 7 and rounded off to the next integer.
Time Frame: Week 4 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: SBMs per week
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 196
SBMs per week | 4.0 (0.42) | 7.8 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.7, 95% CI [2.9 to 4.6], Standard Error of Mean 0.43 — Means are adjusted for center effects and baseline value

11. Secondary Outcome: Time to the First SBM Following the First Dose of Study Medication (SM)
Description: The time to the first SBM following the first dose of SM was captured by the eDiary. The time was censored by the time of intake of rescue medication (RM), the time of premature discontinuation or the end of treatment whatever was minimal.
Time Frame: Time of first dose of SM up to 4 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 114 | 235
Hours | 19 [16 to 25] | 12 [11 to 12]
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; The log-rank test was used to calculate the p-value and to test for differences between the treatment groups; Test type: Superiority or Other; p < 0.0001, Log Rank

12. Secondary Outcome: Number of Participants With an Increase of at Least 1 in the Mean Number of CSBMs Per Week Over the 4 Weeks Treatment Period Compared to Baseline
Time Frame: Baseline and 4 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants | 47 | 196
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 2.04, 95% CI [1.62 to 2.57] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

13. Secondary Outcome: Number of Participants With an Increase of at Least 1 CSBM at Week 1 Compared to Baseline
Time Frame: Baseline and week 1 in treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants | 57 | 204
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 1.75, 95% CI [1.44 to 2.13] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

14. Secondary Outcome: Number of Participants With an Increase of at Least 1 CSBM at Week 2 Compared to Baseline
Time Frame: Baseline and week 2 in treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 115 | 229
Participants | 43 | 178
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 2.08, 95% CI [1.62 to 2.66] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

15. Secondary Outcome: Number of Participants With an Increase of at Least 1 CSBM at Week 3 Compared to Baseline
Time Frame: Baseline and week 3 in treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 113 | 213
Participants | 51 | 163
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 1.70, 95% CI [1.37 to 2.11] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

16. Secondary Outcome: Number of Participants With an Increase of at Least 1 CSBM at Week 4 Compared to Baseline
Time Frame: Baseline and week 4 in treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 196
Participants | 52 | 148
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 1.52, 95% CI [1.24 to 1.88] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

17. Secondary Outcome: Number of Participants With a Mean of at Least 1 CSBM a Day Over the 4 Weeks Treatment Period
Time Frame: 4 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants | 2 | 70
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 17.13, 95% CI [4.28 to 68.66] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

18. Secondary Outcome: Number of Participants With a Mean of at Least 3 CSBMs a Week Over the 4 Weeks Treatment Period
Time Frame: 4 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants | 32 | 161
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 2.46, 95% CI [1.81 to 3.35] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

19. Secondary Outcome: Number of Premature Withdrawals Over the 4 Weeks Treatment Period
Time Frame: 4 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants | 10 | 51
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.0025, Fisher Exact; Odds Ratio (OR) = 2.50, 95% CI [1.32 to 4.74] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

20. Secondary Outcome: Number of Premature Withdrawals at Week 1 in the Treatment Period
Time Frame: Week 1 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants | 3 | 25
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.0105, Fisher Exact; Odds Ratio (OR) = 4.08, 95% CI [1.26 to 13.24] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

21. Secondary Outcome: Number of Premature Withdrawals at Week 2 in the Treatment Period
Time Frame: Week 2 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 115 | 229
Participants | 3 | 11
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.4002, Fisher Exact; Odds Ratio (OR) = 1.84, 95% CI [0.52 to 6.47] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

22. Secondary Outcome: Number of Premature Withdrawals at Week 3 in the Treatment Period
Time Frame: Week 3 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 113 | 214
Participants | 4 | 9
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Odds Ratio (OR) = 1.19, 95% CI [0.37 to 3.77] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

23. Secondary Outcome: Number of Premature Withdrawals at Week 4 in the Treatment Period
Time Frame: Week 4 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 196
Participants | 0 | 6
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.0951, Fisher Exact

24. Secondary Outcome: Number of Participants Using Rescue Medication Over the 4 Weeks Treatment Period
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants | 21 | 8
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Odds Ratio (OR) = 0.19, 95% CI [0.09 to 0.41] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

25. Secondary Outcome: Number of Participants Using Rescue Medication at Week 1 in the Treatment Period
Time Frame: Week 1 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants | 2 | 1
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.2524, Fisher Exact; Odds Ratio (OR) = 0.24, 95% CI [0.02 to 2.67] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

26. Secondary Outcome: Number of Participants Using Rescue Medication at Week 2 in the Treatment Period
Time Frame: Week 2 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 115 | 229
Participants | 10 | 4
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.0035, Fisher Exact; Odds Ratio (OR) = 0.20, 95% CI [0.06 to 0.63] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

27. Secondary Outcome: Number of Participants Using Rescue Medication at Week 3 in the Treatment Period
Time Frame: Week 3 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 113 | 213
Participants | 9 | 1
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.0004, Fisher Exact; Odds Ratio (OR) = 0.06, 95% CI [0.01 to 0.46] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

28. Secondary Outcome: Number of Participants Using Rescue Medication at Week 4 in the Treatment Period
Time Frame: Week 4 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 196
Participants | 12 | 6
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.0086, Fisher Exact; Odds Ratio (OR) = 0.27, 95% CI [0.10 to 0.69] — OR: Bisacodyl / Placebo; The exact 95% confidence interval (CI) by Clopper and Pearson is presented

29. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Straining' at Week 1
Description: The score on a 5-point ordinal verbal rating scale from 0 (absent) to 4 (very severe) specifying patient's symptom assessment associated with each bowel movement was averaged over the day and then averaged over the days in the corresponding week.
Time Frame: Baseline and week 1 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 222
Score on a scale | -0.3 (0.08) | -1.3 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.0, 95% CI [-1.2 to -0.9], Standard Error of Mean 0.08 — Means are adjusted for center effects and baseline value

30. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Straining' at Week 2
Description: as for outcome 29
Time Frame: Baseline and week 2 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 204
Score on a scale | -0.1 (0.09) | -1.1 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.0, 95% CI [-1.2 to -0.8], Standard Error of Mean 0.09 — Means are adjusted for center effects and baseline value

31. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Straining' at Week 3
Description: as for outcome 29
Time Frame: Baseline and week 3 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 100 | 190
Score on a scale | -0.3 (0.09) | -1.3 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.0, 95% CI [-1.1 to -0.8], Standard Error of Mean 0.10 — Means are adjusted for center effects and baseline value

32. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Straining' at Week 4
Description: as for outcome 29
Time Frame: Baseline and week 4 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 96 | 178
Score on a scale | -0.5 (0.10) | -1.2 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI [-0.9 to -0.5], Standard Error of Mean 0.10 — Means are adjusted for center effects and baseline value

33. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Stool Quality' at Week 1
Description: The score on the 7-point Bristol Stool Form Scale from Type 1 (hard, lumpy stool) to Type 7 (watery stool) specifying patient's symptom assessment associated with each bowel movement was averaged over the day and then averaged over the days in the corresponding week.
Time Frame: Baseline and week 1 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 222
Score on a scale | 0.4 (0.13) | 3.0 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.6, 95% CI [2.4 to 2.9], Standard Error of Mean 0.14 — Means are adjusted for center effects and baseline value

34. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Stool Quality' at Week 2
Description: as for outcome 33
Time Frame: Baseline and week 2 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 204
Score on a scale | 0.2 (0.15) | 2.7 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.4, 95% CI [2.1 to 2.7], Standard Error of Mean 0.14 — Means are adjusted for center effects and baseline value

35. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Stool Quality' at Week 3
Description: as for outcome 33
Time Frame: Baseline and week 3 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 100 | 190
Score on a scale | 0.5 (0.14) | 2.8 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.3, 95% CI [2.0 to 2.5], Standard Error of Mean 0.15 — Means are adjusted for center effects and baseline value

36. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Stool Quality' at Week 4
Description: as for outcome 33
Time Frame: Baseline and week 4 in treatment period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 96 | 178
Score on a scale | 0.6 (0.16) | 2.6 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.0, 95% CI [1.7 to 2.3], Standard Error of Mean 0.16 — Means are adjusted for center effects and baseline value

37. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Sensation of Incomplete Evacuation' at Week 1
Description: The score on a 2-point ordinal verbal rating scale from 0 (no) to 1 (yes) specifying patient's symptom assessment associated with each bowel movement was averaged over the day and then averaged over the days in the corresponding week.
Time Frame: Baseline and week 1 in treatment period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 115 | 232
Score on a scale | -0.0 (0.05) | -0.2 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI [-0.3 to -0.1], Standard Error of Mean 0.05 — Means are adjusted for center effects and baseline value

38. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Sensation of Incomplete Evacuation' at Week 2
Description: as for outcome 37
Time Frame: Baseline and week 2 in treatment period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 113 | 220
Score on a scale | -0.0 (0.05) | -0.2 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI [-0.3 to -0.1], Standard Error of Mean 0.05 — Means are adjusted for center effects and baseline value

39. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Sensation of Incomplete Evacuation' at Week 3
Description: as for outcome 37
Time Frame: Baseline and week 3 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 107 | 201
Score on a scale | -0.1 (0.05) | -0.2 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.0127, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI [-0.2 to -0.0], Standard Error of Mean 0.06 — Means are adjusted for center effects and baseline value

40. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Sensation of Incomplete Evacuation' at Week 4
Description: as for outcome 37
Time Frame: Baseline and week 4 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 104 | 188
Score on a scale | -0.1 (0.06) | -0.2 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.0064, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI [-0.3 to -0.0], Standard Error of Mean 0.06 — Means are adjusted for center effects and baseline value

41. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Anorectal Obstructions/Blockade' at Week 1
Description: as for outcome 29
Time Frame: Baseline and week 1 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 222
Score on a scale | -0.1 (0.08) | -0.9 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI [-0.9 to -0.6], Standard Error of Mean 0.08 — Means are adjusted for center effects and baseline value

42. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Anorectal Obstructions/Blockade' at Week 2
Description: as for outcome 29
Time Frame: Baseline and week 2 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 204
Score on a scale | -0.1 (0.09) | -0.9 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI [-1.0 to -0.6], Standard Error of Mean 0.09 — Means are adjusted for center effects and baseline value

43. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Anorectal Obstructions/Blockade' at Week 3
Description: as for outcome 29
Time Frame: Baseline and week 3 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 100 | 190
Score on a scale | -0.1 (0.08) | -0.9 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI [-0.9 to -0.5], Standard Error of Mean 0.09 — Means are adjusted for center effects and baseline value

44. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Anorectal Obstructions/Blockade' at Week 4
Description: as for outcome 29
Time Frame: Baseline and week 4 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 96 | 178
Score on a scale | -0.1 (0.09) | -0.8 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI [-0.8 to -0.5], Standard Error of Mean 0.09 — Means are adjusted for center effects and baseline value

45. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Manual Manoeuvre' at Week 1
Description: as for outcome 37
Time Frame: Baseline and week 1 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 222
Score on a scale | -0.0 (0.03) | -0.2 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI [-0.2 to -0.1], Standard Error of Mean 0.03 — Means are adjusted for center effects and baseline value

46. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Manual Manoeuvre' at Week 2
Description: as for outcome 37
Time Frame: Baseline and week 2 in treatment period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 105 | 204
Score on a scale | 0.0 (0.04) | -0.2 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI [-0.3 to -0.1], Standard Error of Mean 0.04 — Means are adjusted for center effects and baseline value

47. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Manual Manoeuvre' at Week 3
Description: as for outcome 37
Time Frame: Baseline and week 3 in treatment period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 100 | 190
Score on a scale | -0.0 (0.03) | -0.2 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI [-0.2 to -0.1], Standard Error of Mean 0.04 — Means are adjusted for center effects and baseline value

48. Secondary Outcome: Change From Baseline in the Mean Score for Constipation Symptom 'Manual Manoeuvre' at Week 4
Description: as for outcome 37
Time Frame: Baseline and week 4 in treatment period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 96 | 178
Score on a scale | -0.1 (0.04) | -0.2 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.0018, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI [-0.2 to -0.0], Standard Error of Mean 0.04 — Means are adjusted for center effects and baseline value

49. Secondary Outcome: Number of Participants With Improved, Unchanged or Worsened Overall Satisfaction With Bowel Habits at Week 1 in the Treatment Period in Comparison to Baseline
Description: Improved / unchanged / worsened overall satisfaction is a decreased / unchanged / increased score on a 5-point ordinal VRS: 0 (A very great deal satisfied) to 4 (Not at all satisfied) at the corresponding week in comparison to baseline
Time Frame: Baseline and week 1 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 112 | 224
Participants
  Improved overall satisfaction | 44 | 153
  Unchanged overall satisfaction | 46 | 45
  Worsened overall satisfaction | 22 | 26
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

50. Secondary Outcome: Number of Participants With Improved, Unchanged or Worsened Overall Satisfaction With Bowel Habits at Week 2 in the Treatment Period in Comparison to Baseline
Description: as for outcome 49
Time Frame: Baseline and week 2 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 111 | 212
Participants
  Improved overall satisfaction | 41 | 163
  Unchanged overall satisfaction | 48 | 37
  Worsened overall satisfaction | 22 | 12
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

51. Secondary Outcome: Number of Participants With Improved, Unchanged or Worsened Overall Satisfaction With Bowel Habits at Week 3 in the Treatment Period in Comparison to Baseline
Description: as for outcome 49
Time Frame: Baseline and week 3 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 104 | 195
Participants
  Improved overall satisfaction | 44 | 153
  Unchanged overall satisfaction | 43 | 31
  Worsened overall satisfaction | 17 | 11
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

52. Secondary Outcome: Number of Participants With Improved, Unchanged or Worsened Overall Satisfaction With Bowel Habits at Week 4 in the Treatment Period in Comparison to Baseline
Description: as for outcome 49
Time Frame: Baseline and week 4 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 98 | 175
Participants
  Improved overall satisfaction | 37 | 135
  Unchanged overall satisfaction | 47 | 32
  Worsened overall satisfaction | 14 | 8
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

53. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Constipation at Week 1 in the Treatment Period in Comparison to Baseline
Description: Reduced / unchanged / increased bothersomeness of constipation is a decreased / unchanged / increased score on a 5-point ordinal VRS: 0 (Not at all bothersome) to 4 (A very great deal bothersome) at the corresponding week in comparison to baseline
Time Frame: Baseline and week 1 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 112 | 224
Participants
  Reduced bothersomeness | 36 | 168
  Unchanged bothersomeness | 51 | 46
  Increased bothersomeness | 25 | 10
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

54. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Constipation at Week 2 in the Treatment Period in Comparison to Baseline
Description: as for outcome 53
Time Frame: Baseline and week 2 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 111 | 212
Participants
  Reduced bothersomeness | 35 | 160
  Unchanged bothersomeness | 45 | 36
  Increased bothersomeness | 31 | 16
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

55. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Constipation at Week 3 in the Treatment Period in Comparison to Baseline
Description: as for outcome 53
Time Frame: Baseline and week 3 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 104 | 195
Participants
  Reduced bothersomeness | 39 | 147
  Unchanged bothersomeness | 41 | 30
  Increased bothersomeness | 24 | 18
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

56. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Constipation at Week 4 in the Treatment Period in Comparison to Baseline
Description: as for outcome 53
Time Frame: Baseline and week 4 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 98 | 175
Participants
  Reduced bothersomeness | 30 | 125
  Unchanged bothersomeness | 47 | 35
  Increased bothersomeness | 21 | 15
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

57. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Abdominal Bloating at Week 1 in the Treatment Period in Comparison to Baseline
Description: Reduced / unchanged / increased bothersomeness of abdominal bloating is a decreased / unchanged / increased score on a 5-point ordinal VRS: 0 (Not at all bothersome) to 4 (A very great deal bothersome) at the corresponding week in comparison to baseline
Time Frame: Baseline and week 1 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 112 | 224
Participants
  Reduced bothersomeness | 33 | 136
  Unchanged bothersomeness | 47 | 59
  Increased bothersomeness | 32 | 29
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

58. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Abdominal Bloating at Week 2 in the Treatment Period in Comparison to Baseline
Description: as for outcome 57
Time Frame: Baseline and week 2 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 111 | 212
Participants
  Reduced bothersomeness | 31 | 142
  Unchanged bothersomeness | 46 | 43
  Increased bothersomeness | 34 | 27
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

59. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Abdominal Bloating at Week 3 in the Treatment Period in Comparison to Baseline
Description: as for outcome 57
Time Frame: Baseline and week 3 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 104 | 195
Participants
  Reduced bothersomeness | 27 | 129
  Unchanged bothersomeness | 45 | 49
  Increased bothersomeness | 32 | 17
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

60. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Abdominal Bloating at Week 4 in the Treatment Period in Comparison to Baseline
Description: as for outcome 57
Time Frame: Baseline and week 4 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 98 | 175
Participants
  Reduced bothersomeness | 25 | 107
  Unchanged bothersomeness | 46 | 49
  Increased bothersomeness | 27 | 19
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

61. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Abdominal Discomfort at Week 1 in the Treatment Period in Comparison to Baseline
Description: Reduced / unchanged / increased bothersomeness of abdominal discomfort is a decreased / unchanged / increased score on a 5-point ordinal VRS: 0 (Not at all bothersome) to 4 (A very great deal bothersome) at the corresponding week in comparison to baseline
Time Frame: Baseline and week 1 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 112 | 224
Participants
  Reduced bothersomeness | 37 | 93
  Unchanged bothersomeness | 46 | 62
  Increased bothersomeness | 29 | 69
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.6773, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

62. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Abdominal Discomfort at Week 2 in the Treatment Period in Comparison to Baseline
Description: as for outcome 61
Time Frame: Baseline and week 2 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 111 | 212
Participants
  Reduced bothersomeness | 29 | 104
  Unchanged bothersomeness | 49 | 67
  Increased bothersomeness | 33 | 41
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

63. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Abdominal Discomfort at Week 3 in the Treatment Period in Comparison to Baseline
Description: as for outcome 61
Time Frame: Baseline and week 3 in the treatment period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 104 | 195
Participants
  Reduced bothersomeness | 34 | 101
  Unchanged bothersomeness | 33 | 63
  Increased bothersomeness | 37 | 31
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

64. Secondary Outcome: Number of Participants With Reduced, Unchanged or Increased Bothersomeness With Abdominal Discomfort at Week 4 in the Treatment Period in Comparison to Baseline
Description: as for outcome 61
Time Frame: Baseline and week 4 in the treatment period
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 98 | 175
Participants
  Reduced bothersomeness | 31 | 97
  Unchanged bothersomeness | 36 | 46
  Increased bothersomeness | 31 | 32
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for baseline

65. Secondary Outcome: Number of Participants With Respect to the Final Global Assessment of Efficacy by the Investigator
Description: Final global assessment scale range: 1 (good) to 4 (bad), ordinal
Time Frame: 4 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants
  Good | 26 | 156
  Satisfactory | 37 | 59
  Not satisfactory | 30 | 18
  Bad | 24 | 6
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank sum test — Exact p-value

66. Secondary Outcome: Number of Participants With Respect to the Final Global Assessment of Efficacy by the Patient
Description: Final global assessment scale range: 1 (good) to 4 (bad), ordinal
Time Frame: 4 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants
  Good | 23 | 132
  Satisfactory | 35 | 58
  Not satisfactory | 40 | 27
  Bad | 19 | 22
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank sum test — Exact p-value

67. Secondary Outcome: Number of Participants With Respect to the Final Global Assessment of Tolerability by the Investigator
Description: Final global assessment scale range: 1 (good) to 4 (bad), ordinal
Time Frame: 4 weeks
Population: Treated patients ( = All randomised patients, who took at least one dose of trial medication), who provided data for the underlying outcome measure
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants
  Good | 75 | 85
  Satisfactory | 31 | 84
  Not satisfactory | 10 | 43
  Bad | 1 | 27
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank sum test — Exact p-value

68. Secondary Outcome: Number of Participants With Respect to the Final Global Assessment of Tolerability by the Patient
Description: Final global assessment scale range: 1 (good) to 4 (bad), ordinal
Time Frame: 4 weeks
Population: as for outcome 67
Measure: Number; unit: Participants
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Participants
  Good | 38 | 125
  Satisfactory | 50 | 65
  Not satisfactory | 19 | 22
  Bad | 10 | 27
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Test type: Superiority or Other; p = 0.0058, Wilcoxon rank sum test — Exact p-value

69. Secondary Outcome: Change From Baseline in the SF-36 Dimension 'Physical Functioning'
Description: The dimension is a sum of 10 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
Time Frame: Baseline and 4 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -0.6 (1.92) | -0.0 (1.55)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.7980, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.5, 95% CI [-3.4 to 4.5], Standard Error of Mean 2.01 — Means are adjusted for center effects and baseline value

70. Secondary Outcome: Change From Baseline in the SF-36 Dimension 'Role Limitation Due to Physical Problems'
Description: The dimension is a sum of 4 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
Time Frame: Baseline and 4 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -0.2 (1.96) | 0.9 (1.58)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.6129, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.0, 95% CI [-3.0 to 5.1], Standard Error of Mean 2.05 — Means are adjusted for center effects and baseline value

71. Secondary Outcome: Change From Baseline in the SF-36 Dimension 'Bodily Pain'
Description: The dimension is a sum of 2 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
Time Frame: Baseline and 4 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -2.3 (2.21) | -0.2 (1.78)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.3567, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.1, 95% CI [-2.4 to 6.7], Standard Error of Mean 2.31 — Means are adjusted for center effects and baseline value

72. Secondary Outcome: Change From Baseline in the SF-36 Dimension 'General Health'
Description: The dimension is a sum of 5 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
Time Frame: Baseline and 4 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -1.3 (1.28) | 0.7 (1.03)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.1407, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.0, 95% CI [-0.7 to 4.6], Standard Error of Mean 1.34 — Means are adjusted for center effects and baseline value

73. Secondary Outcome: Change From Baseline in the SF-36 Dimension 'Vitality'
Description: as for outcome 70
Time Frame: Baseline and 4 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -1.6 (1.66) | 2.7 (1.34)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.0130, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.3, 95% CI [0.9 to 7.7], Standard Error of Mean 1.74 — Means are adjusted for center effects and baseline value

74. Secondary Outcome: Change From Baseline in the SF-36 Dimension 'Social Functioning'
Description: as for outcome 71
Time Frame: Baseline and 4 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -2.6 (2.04) | -1.5 (1.64)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.5849, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI [-3.0 to 5.3], Standard Error of Mean 2.14 — Means are adjusted for center effects and baseline value

75. Secondary Outcome: Change From Baseline in the SF-36 Dimension 'Role Limitation Due to Emotional Problems'
Description: The dimension is a sum of 3 single items and then transferred to a scale ranging from 0 to 100. Single item scores are inverted, if applicable, to ensure that a higher score indicates a better health.
Time Frame: Baseline and 4 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -0.5 (1.85) | 0.1 (1.49)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.7543, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI [-3.2 to 4.4], Standard Error of Mean 1.94 — Means are adjusted for center effects and baseline value

76. Secondary Outcome: Change From Baseline in the SF-36 Dimension 'Mental Health'
Description: as for outcome 72
Time Frame: Baseline and 4 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -2.9 (1.52) | 0.6 (1.22)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.0273, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.5, 95% CI [0.4 to 6.6], Standard Error of Mean 1.58 — Means are adjusted for center effects and baseline value

77. Secondary Outcome: Change From Baseline in the SF-36 Mental Component Scale (MCS)
Description: The MCS is a summary scale of the dimensions vitality, social functioning, role-emotional, and mental health. The component scale is norm-based to a standard population. A higher score indicates a better health.
Time Frame: Baseline and 4 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -1.0 (0.82) | 0.3 (0.66)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.1290, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.3, 95% CI [-0.4 to 3.0], Standard Error of Mean 0.87 — Means are adjusted for center effects and baseline value

78. Secondary Outcome: Change From Baseline in the SF-36 Physical Component Scale (PCS)
Description: The PCS is a summary scale of the subscales physical functioning, role-physical, bodily pain, and general health. The component scale is norm-based to a standard population. A higher score indicates a better health.
Time Frame: Baseline and 4 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -0.4 (0.66) | 0.3 (0.53)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.3780, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI [-0.8 to 2.0], Standard Error of Mean 0.70 — Means are adjusted for center effects and baseline value

79. Secondary Outcome: Change From Baseline in the PAC-QoL Subscale 'Worries and Concerns'
Description: The PAC-QoL is a 28-item (5-point Likert scale ranging from 0 (none of the time or not at all) to 4 (all of the time or extremely). Single item scores are inverted, if applicable, to ensure that a lower score indicates a better QoL
Time Frame: Baseline and 4 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -0.1 (0.07) | -0.6 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI [-0.6 to -0.3], Standard Error of Mean 0.08 — Means are adjusted for center effects and baseline value

80. Secondary Outcome: Change From Baseline in the PAC-QoL Subscale 'Physical Discomfort'
Description: as for outcome 79
Time Frame: Baseline and 4 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -0.2 (0.09) | -1.0 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI [-1.0 to -0.7], Standard Error of Mean 0.09 — Means are adjusted for center effects and baseline value

81. Secondary Outcome: Change From Baseline in the PAC-QoL Subscale 'Psychosocial Discomfort'
Description: as for outcome 79
Time Frame: Baseline and 4 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -0.1 (0.07) | -0.3 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p = 0.0070, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI [-0.3 to -0.1], Standard Error of Mean 0.07 — Means are adjusted for center effects and baseline value

82. Secondary Outcome: Change From Baseline in the PAC-QoL Subscale 'Satisfaction'
Description: as for outcome 79
Time Frame: Baseline and 4 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -0.2 (0.12) | -1.4 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.2, 95% CI [-1.5 to -1.0], Standard Error of Mean 0.13 — Means are adjusted for center effects and baseline value

83. Secondary Outcome: Change From Baseline in the PAC-QoL Overall Score
Description: as for outcome 79
Time Frame: Baseline and 4 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 117 | 239
Score on a scale | -0.1 (0.08) | -0.8 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Bisacodyl; Analysis of covariance (ANCOVA) including centre as fixed effect and baseline as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI [-0.8 to -0.5], Standard Error of Mean 0.08 — Means are adjusted for center effects and baseline value

84. Secondary Outcome: Change From Baseline for Sodium (Normalized Value)
Description: Normalized value: the reported laboratory value is converted by linear transformation to a preferred unit and then linear-transformed with respect to the standard reference range
Time Frame: Baseline and 4 weeks
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 114 | 235
mmol/L | -0 (3) | -0 (3)

85. Secondary Outcome: Change From Baseline for Potassium (Normalized Value)
Description: as for outcome 84
Time Frame: Baseline and 4 weeks
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 114 | 235
mmol/L | 0.0 (0.3) | -0.0 (0.3)

86. Secondary Outcome: Change From Baseline for Chloride (Normalized Value)
Description: as for outcome 84
Time Frame: Baseline and 4 weeks
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Bisacodyl
Number analyzed (Participants) | 114 | 235
mmol/L | 0 (3) | 0 (3)

ADVERSE EVENTS:
Time Frame: 4 Weeks
Arm/Group | Placebo | Bisacodyl
Serious Adverse Events (participants affected / at risk) | 2/121 | 1/247
Other Adverse Events (participants affected / at risk) | 14/121 | 159/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=121) | Bisacodyl (N=247)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Chest pain (General disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=121) | Bisacodyl (N=247)
Diarrhoea (Gastrointestinal disorders) | 2 | 132
Abdominal pain (Gastrointestinal disorders) | 3 | 61
Abdominal pain upper (Gastrointestinal disorders) | 3 | 19
Headache (Nervous system disorders) | 7 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.